CLINICAL TRIAL: NCT00772109
Title: Lot Consistency, Immunogenicity, and Safety Study of Three Lots of Fluzone Vaccine Administered by Intradermal Route in Comparison With Standard Fluzone® Administered Intramuscularly in Adult Subjects Aged 18 to 64 Years
Brief Title: Study of Fluzone Vaccine Administered by Intradermal Route in Comparison With Standard Fluzone® in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FID31
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Orthomyxoviridae Infection; Influenza; Myxovirus Infection
Keywords: Influenza; Orthomyxoviruses; Inactivated Split-virion influenza vaccine; Fluzone®; Adults
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fluzone Intradermal Vaccine Lot 1 (Experimental): Participants will receive a dose of Influenza intradermal vaccine Lot 1
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B
- Fluzone Intradermal Vaccine Lot 2 (Experimental): Participants will receive a dose of Influenza intradermal vaccine Lot 2
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B
- Fluzone Intradermal Vaccine Lot 3 (Experimental): Participants will receive a dose of Influenza intradermal vaccine Lot 3
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B
- Fluzone Intramuscular Vaccine (Active Comparator): Participants will receive a dose of influenza intramuscular vaccine
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B

INTERVENTIONS:
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.1 mL, Intradermal
  Arms: Fluzone Intradermal Vaccine Lot 1
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.1 mL, Intradermal
  Arms: Fluzone Intradermal Vaccine Lot 2
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.1 mL, Intradermal
  Arms: Fluzone Intradermal Vaccine Lot 3
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Fluzone Intramuscular Vaccine

SUMMARY:
This study is designed to test lot consistency of three different manufacturing lots and to generate safety and immunogenicity data of the investigational vaccine administered via the ID route.

Primary Objective:

* To demonstrate lot consistency of the Fluzone ID manufacturing process.
* To provide information concerning the immune response of Fluzone ID.

Secondary Objectives:

Safety

* To describe the safety profile of subjects who receive of Fluzone ID.

DETAILED DESCRIPTION:
Three lots of the investigational Fluzone vaccine with the 2008/2009 Northern Hemisphere formulation will be administered intradermally (ID) using the Becton Dickinson Micro Injection System.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 to 64 years on the day of vaccination.
* Informed consent form signed and dated.
* Able to attend all scheduled visits and to comply with all trial procedures.
* For women of child bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to vaccination, until at least 4 weeks after vaccination.

Exclusion Criteria :

* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances.
* For a woman of child-bearing potential: known pregnancy or positive serum/urine pregnancy test.
* Breast-feeding woman.
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the four weeks preceding the trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Chronic illness, at a stage that could interfere with trial conduct or completion, in the opinion of the investigator.
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures.
* Receipt of blood or blood-derived products in the past 3 months that might interfere with the assessment of immune response.
* Receipt of any vaccination in the 4 weeks preceding the trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination.
* Previous vaccination against influenza in the past 6 months with the trial vaccine or another vaccine.
* Thrombocytopenia or bleeding disorder in the 3 weeks preceding inclusion.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* Neoplastic disease or any hematologic malignancy, (except localized skin or prostate cancer that is stable at the time of vaccination in the absence of therapy, and subjects who have a history of neoplastic disease and who have been disease free for >=5 years).
* Personal or family history of Guillain-Barré Syndrome.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4292 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (45):
- United States (43):
  - Hoover, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Fountain Valley, California
  - San Diego, California
  - Milford, Connecticut
  - Melbourne, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Iowa City, Iowa
  - Wichita, Kansas
  - Lexington, Kentucky
  - Madisonville, Kentucky
  - Rockville, Maryland
  - Kansas City, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Binghamton, New York
  - Endwell, New York
  - Rochester, New York
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Allentown, Pennsylvania
  - Bensalem, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Galveston, Texas
  - San Angelo, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Seattle, Washington
  - Marshfield, Wisconsin
- Puerto Rico (2):
  - Castellana Gardens, Carolina
  - San Juan

REFERENCES:
- [Derived] Gorse GJ, Falsey AR, Fling JA, Poling TL, Strout CB, Tsang PH. Intradermally-administered influenza virus vaccine is safe and immunogenic in healthy adults 18-64 years of age. Vaccine. 2013 May 1;31(19):2358-65. doi: 10.1016/j.vaccine.2013.03.008. Epub 2013 Mar 13. PMID 23499604
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 13 through 30 October 2008 in 50 clinics in the US.
Pre-assignment Details: A total of 4276 of the 4292 participants that met the inclusion and exclusion criteria enrolled were vaccinated.
Groups:
- Fluzone Intradermal (ID) Vaccine Lot 1: Participants received a dose of Fluzone Intradermal (ID) vaccine Lot 1 on Day 0
- Fluzone Intradermal (ID) Vaccine Lot 2: Participants received a dose of Fluzone Intradermal (ID) vaccine Lot 2 on Day 0
- Fluzone Intradermal (ID) Vaccine Lot 3: Participants received a dose of Fluzone Intradermal (ID) vaccine Lot 3 on Day 0
- Fluzone Intramuscular (IM) Vaccine: Participants received a dose of Fluzone Intramuscular (IM) vaccine on Day 0
Period: Overall Study
Arm/Group | Fluzone Intradermal (ID) Vaccine Lot 1 | Fluzone Intradermal (ID) Vaccine Lot 2 | Fluzone Intradermal (ID) Vaccine Lot 3 | Fluzone Intramuscular (IM) Vaccine
Started | 956 | 953 | 955 | 1428
Completed | 935 | 934 | 936 | 1397
Not Completed | 21 | 19 | 19 | 31
Not completed — Serious adverse event | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 5 | 8 | 7 | 6
Not completed — Lost to Follow-up | 7 | 3 | 5 | 9
Not completed — Withdrawal by Subject | 8 | 8 | 6 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone Intradermal (ID) Vaccine Lot 1 | Fluzone Intradermal (ID) Vaccine Lot 2 | Fluzone Intradermal (ID) Vaccine Lot 3 | Fluzone Intramuscular (IM) Vaccine | Total
Number analyzed (Participants) | 956 | 953 | 955 | 1428 | 4292
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 956 | 953 | 955 | 1428 | 4292
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (13.41) | 42.8 (13.33) | 42.2 (13.78) | 42.5 (13.55) | 42.5 (13.5175)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 611 | 619 | 594 | 899 | 2723
  Male | 345 | 334 | 361 | 529 | 1569
Region of Enrollment [Number; unit: Participants]
  United States | 956 | 953 | 955 | 1428 | 4292

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) at Baseline and Post-vaccination With Either Fluzone Intradermal or Fluzone Intramuscular Vaccines
Description: The serological determinations of anti influenza antibodies was by Hemagglutination Inhibition (HAI) assay
Time Frame: Baseline (Day 0) and 28 Days post-vaccination
Population: Geometric Mean Titers (GMTs) were analyzed in the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluzone Intradermal (ID) Vaccine Lot 1 | Fluzone Intradermal (ID) Vaccine Lot 2 | Fluzone Intradermal (ID) Vaccine Lot 3 | Fluzone Intramuscular (IM) Vaccine
Number analyzed (Participants) | 863 | 856 | 860 | 1286
Titer
  A/H1N1 (Pre-vaccination, N = 863, 856, 860, 1285) | 23.50 [21.58 to 25.60] | 25.27 [23.16 to 27.58] | 25.29 [23.20 to 27.56] | 24.84 [23.16 to 26.65]
  A/H1N1 (Post-vaccination, N = 863, 855, 861, 1283) | 188.56 [172.67 to 205.92] | 185.59 [169.81 to 202.83] | 206.10 [188.53 to 225.31] | 178.30 [166.36 to 191.11]
  A/H3N2 (Pre-vaccination, N = 862, 853, 860, 1286) | 18.77 [17.29 to 20.38] | 20.56 [18.89 to 22.38] | 18.37 [16.88 to 19.99] | 19.99 [18.65 to 21.43]
  A/H3N2 (Post-vaccination, N = 862, 853, 860, 1284) | 260.46 [235.49 to 288.09] | 234.03 [212.13 to 258.21] | 246.06 [222.65 to 271.93] | 230.71 [213.75 to 249.03]
  B (Pre-vaccination, N = 862, 855, 860, 1286) | 23.77 [22.03 to 25.63] | 25.59 [23.69 to 27.64] | 24.24 [22.51 to 26.10] | 25.05 [23.53 to 26.68]
  B (Post-vaccination, N = 861, 856, 860, 1285) | 103.72 [96.61 to 111.35] | 102.91 [95.88 to 110.46] | 100.82 [93.95 to 108.20] | 126.91 [119.70 to 134.56]

2. Primary Outcome: Percentage of Participants Who Achieved Seroconversion Post-vaccination With Either Fluzone Intradermal or Fluzone Intramuscular Vaccine
Description: The serological determinations of anti influenza antibodies was by Hemagglutination Inhibition (HAI) assay.
  Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and post-vaccination titer of ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and a minimum of four-fold increase 28 days post-vaccination.
Time Frame: 28 Days post-vaccination
Population: Seroprotection was analyzed in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone Intradermal (ID) Vaccine Lot 1 | Fluzone Intradermal (ID) Vaccine Lot 2 | Fluzone Intradermal (ID) Vaccine Lot 3 | Fluzone Intramuscular (IM) Vaccine
Number analyzed (Participants) | 863 | 856 | 860 | 1286
Percentage of Participants
  A/H1N1 Serogroup | 61 | 59 | 63 | 61
  A/H3N2 Serogroup | 76 | 73 | 77 | 75
  B Serogroup | 47 | 45 | 47 | 54

3. Secondary Outcome: Percentage of Participants Who Achieved Seroprotection Pre- and Post-vaccination With Either Fluzone ID or Fluzone IM
Description: The serological determinations of anti influenza antibodies was by Hemagglutination Inhibition (HAI) assay.
  Seroprotection was defined as a HAI antibody titer ≥ 1:40.
Time Frame: Before and 28 Days post-vaccination
Population: 4-Fold increase in antibody levels were analyzed in h per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone Intradermal (ID) Vaccine Lot 1 | Fluzone Intradermal (ID) Vaccine Lot 2 | Fluzone Intradermal (ID) Vaccine Lot 3 | Fluzone Intramuscular (IM) Vaccine
Number analyzed (Participants) | 863 | 857 | 861 | 1287
Percentage of Participants
  A/H1N1 Serogroup (Pre-vaccination) | 39 | 40 | 42 | 39
  A/H1N1 Serogroup (Post-vaccination) | 90 | 90 | 93 | 92
  A/H3N2 Serogroup (Pre-vaccination) | 31 | 32 | 30 | 34
  A/H3N2 Serogroup (Post-vaccination) | 92 | 90 | 91 | 91
  B Serogroup (Pre-vaccination) | 38 | 42 | 40 | 41
  B Serogroup (Post-vaccination) | 88 | 88 | 86 | 89

4. Secondary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reactions, Post Vaccination With Either Fluzone Intradermal or Fluzone Intramuscular Vaccine
Description: Solicited injection site reactions: Ecchymosis, Erythema, Induration, Pain, Pruritus, and Swelling. Solicited systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Shivering.
Time Frame: Day 0 up to 7 Days post vaccination
Population: Safety analysis was on all enrolled and vaccinated participants, intend-to-treat population
Measure: Number; unit: Participants
Arm/Group | Fluzone Intradermal (ID) Vaccine Lot 1 | Fluzone Intradermal (ID) Vaccine Lot 2 | Fluzone Intradermal (ID) Vaccine Lot 3 | Fluzone Intramuscular (IM) Vaccine
Number analyzed (Participants) | 953 | 951 | 951 | 1421
Participants
  Any Injection Site Ecchymosis | 81 | 82 | 97 | 86
  Grade 3 Injection Site Ecchymosis (≥ 5 cm) | 8 | 2 | 2 | 6
  Any Injection Site Erythema | 716 | 698 | 726 | 184
  Grade 3 Injection Site Erythema (≥ 5 cm) | 125 | 118 | 120 | 13
  Any Injection Site Induration | 554 | 533 | 547 | 139
  Grade 3 Injection Site Induration (≥ 5 cm) | 36 | 19 | 41 | 7
  Any Injection Site Pain | 480 | 449 | 500 | 749
  Grade 3 Injection Site Pain (Incapacitating) | 3 | 6 | 9 | 11
  Any Injection Site Pruritus | 447 | 430 | 438 | 129
  Grade 3 Injection Site Pruritus (Incapacitating) | 13 | 10 | 7 | 0
  Any Injection Site Swelling | 544 | 525 | 519 | 117
  Grade 3 Injection Site Swelling (≥ 5 cm) | 55 | 45 | 52 | 13
  Any Solicited Fever | 29 | 40 | 40 | 36
  Grade 3 Solicited Fever (> 102.2°F) | 2 | 0 | 0 | 3
  Any Solicited Headache | 282 | 279 | 314 | 422
  Gr 3 Solicited Headache- Prevents daily activities | 11 | 16 | 14 | 22
  Any Solicited Malaise | 212 | 202 | 239 | 309
  Grd 3 Solicited Malaise- Prevents daily activities | 19 | 26 | 17 | 25
  Any Solicited Myalgia | 252 | 229 | 260 | 430
  Grd 3 Solicited Myalgia- Prevents daily activities | 13 | 18 | 10 | 19
  Any Solicited Shivering | 71 | 56 | 77 | 87
  Gr 3 Solicited Shivering-Prevents daily activities | 7 | 8 | 6 | 9

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for up to 6 months post-vaccination.
Arm/Group | Fluzone Intradermal (ID) Vaccine Lot 1 | Fluzone Intradermal (ID) Vaccine Lot 2 | Fluzone Intradermal (ID) Vaccine Lot 3 | Fluzone Intramuscular (IM) Vaccine
Serious Adverse Events (participants affected / at risk) | 17/953 | 16/951 | 14/951 | 20/1421
Other Adverse Events (participants affected / at risk) | 716/953 | 698/951 | 726/951 | 749/1421
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone Intradermal (ID) Vaccine Lot 1 (N=953) | Fluzone Intradermal (ID) Vaccine Lot 2 (N=951) | Fluzone Intradermal (ID) Vaccine Lot 3 (N=951) | Fluzone Intramuscular (IM) Vaccine (N=1421)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Non cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsi (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stent occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Fluzone Intradermal (ID) Vaccine Lot 1 (N=953) | Fluzone Intradermal (ID) Vaccine Lot 2 (N=951) | Fluzone Intradermal (ID) Vaccine Lot 3 (N=951) | Fluzone Intramuscular (IM) Vaccine (N=1421)
Injection site ecchymosis (General disorders) | 81/935 (81) | 82/935 (82) | 97/929 (97) | 86/1392 (86)
Injection site erythema (General disorders) | 716/936 (716) | 698/935 (698) | 726/930 (726) | 184/1393 (184)
Injection site induration (General disorders) | 554/934 (554) | 533/935 (533) | 547/929 (547) | 139/1392 (139)
Injection site pain (General disorders) | 480/936 (480) | 449/935 (449) | 500/931 (500) | 749/1394 (749)
Injection site pruritus (General disorders) | 447/936 (447) | 430/935 (430) | 438/931 (438) | 129/1394 (129)
Injection site swelling (General disorders) | 544/934 (544) | 525/935 (525) | 519/929 (519) | 117/1392 (117)
Solicited Headache (Nervous system disorders) | 282/936 (282) | 279/935 (279) | 314/930 (314) | 422/1394 (422)
Solicited Malaise (General disorders) | 212/936 (212) | 202/935 (202) | 239/930 (239) | 309/1394 (309)
Solicited Myalgia (Musculoskeletal and connective tissue disorders) | 252/936 (252) | 229/935 (229) | 260/930 (260) | 430/1394 (430)
Solicited Shivering (Musculoskeletal and connective tissue disorders) | 71/936 (71) | 56/935 (56) | 77/930 (77) | 87/1394 (87)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.